CLINICAL TRIAL: NCT04691362
Title: Study of the Noninferiority of an Oral vs Intravenous Administration of Tranexamic Acid in Total Hip Arthroplasty
Brief Title: Noninferiority Oral Tranexamic Acid vs Intravenous Administration in Total Hip Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Jean François Brichant, Head of Anesthesiology Departement, University of Liege
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 2020-316
Record Dates: First submitted 2020-12-29; First posted 2020-12-31 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Hemorrhage Postoperative; Total Blood Loss; Arthroplasty Complications
MeSH Terms: conditions — Postoperative Hemorrhage; Exsanguination | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blinded randomized controlled trial. Patient, anesthesiologist and surgeon are blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral Tranexamic Acid (Active Comparator): 128 patients scheduled for primary total hip arthroplasty
  Interventions: Drug: Tranexamic Acid Oral Product
- Intravenous Tranexamic Acid (Active Comparator): 128 patients scheduled for primary total hip arthroplasty
  Interventions: Drug: Tranexamic acid injection

INTERVENTIONS:
Drug: Tranexamic Acid Oral Product — Oral administration of 2 grammes tranexamic acid 2 hours before skin incision and 2 grammes oral tranexamic acid 4 hours after first administration
  Arms: Oral Tranexamic Acid
Drug: Tranexamic acid injection — Intravenous administration of 1 gramme tranexamic acid 30 minutes before skin incision and 1 gramme intravenous tranexamic acid 4 hours after first administration
  Arms: Intravenous Tranexamic Acid

SUMMARY:
To find noninferiority relationship between oral and intravenous administration of tranexamic acid on peroperative and postoperative blood loss and serum concentration during primary total hip arthroplasty.

DETAILED DESCRIPTION:
Tranexamic acid is an anti-fibrinolytic drug, recommended in total hip arthroplasty to reduce peroperative and postoperative hemorrhagic complications. The original character of our study lies in the serum dosage of tranexamic acid, allowing to correlate the primary objective (blood loss) with this one. The investigators will focus on the reduction of the risks associated with the administration of intravenous medicines, the economic aspect and the ease of use.

ELIGIBILITY:
Inclusion Criteria:

- ASA physical status 1, 2 and 3 scheduled for primary total hip arthroplasty

Exclusion Criteria:

* Renal failure with serum creatinine level higher than 1,40 mg/dL
* Thromboembolic events in last 12 months before surgery
* Pregnancy
* Congenital or acquired coagulation diseases
* History of gastric surgery that could lead to malabsorption
* Diabetic gastro-paresis

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-12-14 (Actual); Study Completion 2022-12-14 (Actual)

PRIMARY OUTCOMES:
Total blood loss | First 48 hours after surgery
  Peroperative (suction) and postoperative (drainage) total blood loss

SECONDARY OUTCOMES:
Serum concentration of tranexamic acid | 2 hours after oral administration
  Monitoring of serum dosage of tranxemaic acid in randomized subpopulation of each group
Serum concentration of tranexamic acid | 6 hours after oral administration
  Monitoring of serum dosage of tranxemaic acid in randomized subpopulation of each group
Serum concentration of tranexamic acid | 30 minutes after intravenous administration
  Monitoring of serum dosage of tranxemaic acid in randomized subpopulation of each group
Serum concentration of tranexamic acid | 4 hours after intravenous administration
  Monitoring of serum dosage of tranxemaic acid in randomized subpopulation of each group
Serum hemoglobin variation | 24 hours after surgery
  Variation of serum hemoglobin between preoperative and postoperative period
Serum hemoglobin variation | 72 hours after surgery
  Variation of serum hemoglobin between preoperative and postoperative period
Incidence of blood transfusion | 72 hours after surgery
  Incidence of blood transfusion in two groups
Incidence of thromboembolic complications | 72 hours after surgery
  Incidence of thromboembolic complications such as pulmonary embolism or deep venous thrombosis
Length of hospitalisation stay | 1 week after surgery
  Difference between two groups of total hospitalisation days

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Liège, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fillingham YA, Ramkumar DB, Jevsevar DS, Yates AJ, Bini SA, Clarke HD, Schemitsch E, Johnson RL, Memtsoudis SG, Sayeed SA, Sah AP, Della Valle CJ. Tranexamic acid in total joint arthroplasty: the endorsed clinical practice guides of the American Association of Hip and Knee Surgeons, American Society of Regional Anesthesia and Pain Medicine, American Academy of Orthopaedic Surgeons, Hip Society, and Knee Society. Reg Anesth Pain Med. 2019 Jan;44(1):7-11. doi: 10.1136/rapm-2018-000024. No abstract available. PMID 30640647
- [Background] Wu Y, Zeng Y, Hu Q, Li M, Bao X, Zhong J, Shen B. Blood loss and cost-effectiveness of oral vs intravenous tranexamic acid in primary total hip arthroplasty: A randomized clinical trial. Thromb Res. 2018 Nov;171:143-148. doi: 10.1016/j.thromres.2018.10.006. Epub 2018 Oct 6. PMID 30312799
- [Derived] Piette N, Beck F, Carella M, Hans G, Maesen D, Kurth W, Lecoq JP, Bonhomme VL. Oral as compared to intravenous tranexamic acid to limit peri-operative blood loss associated with primary total hip arthroplasty: A randomised noninferiority trial. Eur J Anaesthesiol. 2024 Mar 1;41(3):217-225. doi: 10.1097/EJA.0000000000001950. Epub 2024 Jan 12. PMID 38214552